**ID RCB**: not applicable

Sponsor ID: QS-NIS-G-H-2101

**Title of document: Protocol synopsis** 

Date: 03-OCT-2022 Version: 2.0



## POST MARKET FOLLOW-UP STUDY OF A ROBOTIC DEVICE FOR IMAGE-GUIDED PERCUTANEOUS NEEDLE PLACEMENT IN THE ABDOMEN

| Study title | Post Market Clinical Follow-up study of a robotic device for image-guided percutaneous needle placement in the abdomen |
|---|---|
| Study Number | QS-NIS-G-H-2101 |
| Investigational product | EPIONE® device |
| Investigational product characteristics | The device is a user controlled, stereotactic accessory intended to assist in the planning and manual advancement of needle, as well as in verification of needle position during CT-guided percutaneous ablation procedures. |
| Investigational device administration | The operating principle of the investigational device is the following: pre-interventional CT-scan acquisition, planning with the device's software, needle's insertion according to the predefined planning, acquisition of a per-procedure CT-scan to evaluate the needle(s) placement. |
| Reference therapy/product | N/A |
| Study design | Post Market Clinical Follow-up study (PMCF) |
| | Non-interventional, prospective, non-comparative study |
| Number of sites & country | 1 site in France |
| Sample size | Around 55 patients |
| | Around 55 CT-guided procedures in the abdomen |
| Indication | Percutaneous CT-guided procedures (tumor ablation, biopsy,) in the abdomen (liver, kidney,) |

ID RCB : not applicable

Sponsor ID: QS-NIS-G-H-2101

**Title of document : Protocol synopsis** 

Date: 03-OCT-2022 Version: 2.0



| Primary objective | Evaluation of the technical success of the device |
|---|---|
| Primary endpoint | Number of targets reached; the target is considered to have been reached when the needle is positioned accurately enough to allow the planned procedure to be performed. |
| Secondary<br>objective | Assessment of performance parameters and safety |
| Secondary<br>endpoint | Performance parameters |
| | Safety o Adverse Event(s) (AEs) |
| Patient inclusion/exclusion criteria | Inclusion criteria: 1. Patient is >18 years old, 2. Patient for whom a CT-guided procedure in abdomen has been prescribed and agreed by a multidisciplinary team of radiologists, surgeons and clinicians, 3. Patient with a confirmed non-opposition. Exclusion criteria: 1. Patient unable to undergo general anesthesia, Pregnant or breast-feeding female |
| Visit schedule | Schematic diagram of visit schedule: |
| | Routine Day of the Routine follow-up Routine follow-up pre-intervention intervention visit at 2M Visit at 10M consultation |
| | <ul> <li>Visit 1: initial visit – patient screening (D0-1 month) ≤D≤D0 </li> <li>Review of inclusion and exclusion criteria, presentation of the study and the device (oral and written information for the patient). Paper information</li> </ul> |

**ID RCB**: not applicable

Sponsor ID : QS-NIS-G-H-2101

**Title of document: Protocol synopsis** 

Date: 03-OCT-2022 Version: 2.0



notice and non-opposition forms discussed with the patient allowing them sufficient time to consider the study's implications before deciding whether to participate. Next visit planned (day of the CT-guided intervention).

- <u>Visit 2: inclusion visit procedure day</u>
   D0
- Confirmation of the non-opposition by the investigator,
- Collection of demographic data, tumor data, primary cancer data as well as other medical history. Collection of concomitants pathologies/treatments.
- Patient placed under general anesthesia.
- Acquisition of the pre-interventional CT-guided image for the planning phase.
- Insertion of the needle(s) to the targeted area with the subject device.
- Acquisition of the per-procedure image under CT guidance.
- Validation of the correct positioning of the needle(s).
- Acquisition of the post-interventional CT-guided image.
- Visit 3: post-intervention follow-up visit at 2 months (D0+3 weeks≤D≤D0+3 months)

Acquisition of an image (CT-guided or MRI) of the organ to evaluate ablation site recurrence (local tumor recurrence) and possible AEs.

 Visit 4: post-intervention follow-up visit at 10 months (D0+6 months≤D≤D0+15 months)

Acquisition of an image (CT-guided or MRI) of the organ to evaluate ablation site recurrence (local tumor recurrence) and possible AEs.

Study duration per patient

From patient's information and non-opposition form signature to visit 4. From 6 months to 16 months, depending on the day of patient's non-opposition confirmation and the day of the visit 4.

Study schedule Planned start: Q1 2022
Planned recruitment time: 18 months
Planned last patient out: Q1 2024

Randomization/
No randomization, open label blinding

Non

GCP statement

**DSMB** 

This study will be conducted in compliance with the protocol, the current version of the Declaration of Helsinki, the ICH-GCP and ISO EN 14155 as well as all national legal and regulatory requirements.